CLINICAL TRIAL: NCT05798975
Title: Analysis of Heart Rate Variability After One Session of Aerobic or Resistance Physical Exercise in Controlled Hypertensive Individuals: Randomized Clinical Trial
Brief Title: Analysis of Heart Rate Variability After a Physical Exercise Session
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Diego Silveira da Silva, physical education professor., Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5964/21
Record Dates: First submitted 2023-02-10; First posted 2023-04-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: AE= Aerobic Exercise RE= Resistance Exercise CT= Control (no exercise)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Physical Exercise (Experimental): Cycle ergometer exercise
  Interventions: Other: Resistance Exercise. 1 session of acute exercise; Other: no exercise
- Resistance Physical Exercise (Experimental): Exercise with weights
  Interventions: Other: Aerobic Exercise. 1 session of acute exercise; Other: no exercise
- Control (No Intervention): No exercise. Rest

INTERVENTIONS:
Other: Aerobic Exercise. 1 session of acute exercise — 40 minutes on cycle ergometer, 60% of heart rate reserve
  Arms: Resistance Physical Exercise
Other: Resistance Exercise. 1 session of acute exercise — 2 exercises for lower limbs and 2 for upper limbs with 4 sets of 12 repetitions at 60% 1-RM. 40 minutes
  Arms: Aerobic Physical Exercise
Other: no exercise — Rest
  Arms: Aerobic Physical Exercise; Resistance Physical Exercise

SUMMARY:
Systemic arterial hypertension (SAH) is a multifactorial clinical condition, characterized by sustained elevation of blood pressure levels, contributing to 50% of deaths from cardiovascular disease. The Autonomic Nervous System (ANS) plays a fundamental role in the regulation of Blood Pressure (BP) and is closely associated with Heart Rate (HR). HR changes are called Heart Rate Variability (HRV). In individuals with SAH, HRV indices are reduced compared to normotensive individuals, showing changes in autonomic modulation, thus increasing the risk for cardiovascular events. The objective of this study will be to analyze the Heart Rate Variability in individuals with controlled SAH after a session of aerobic (EA) or resistance (RE) physical exercise.

DETAILED DESCRIPTION:
Controlled hypertensive individuals aged between 30 and 59 years will be selected, for convenience, who use the services of the Instituto de Cardiologia do Rio Grande do Sul. Volunteers will be randomly assigned to an EA session (40 minutes on cycle ergometer, 60% of heart rate reserve) or RE (2 exercises for lower limbs and 2 for upper limbs with 4 sets of 12 repetitions at 60% 1-RM) or control group without exercise. HRV data will be collected by ECG (Wincardio USB - Version 11.1.0.0, MICROMED Biotecnologia Ltda, Brasília - DF - Brazil) during 10 minutes before the exercise session, 10 minutes after the exercise session, 1h and 2h post-session . It is expected to estimate results that may demonstrate clarifications about the impact of a physical exercise session on HRV in controlled hypertensive individuals.

ELIGIBILITY:
Inclusion Criteria:

* Controlled Systemic Alterial Hypertension

Exclusion Criteria:

* Diabetes mellitus;
* heart failure;
* coronary artery disease;
* chronic renal failure;
* body mass index (BMI) ≥ 35 kg/m2;
* smokers;
* individuals with injuries to the upper and lower limbs that make the exercise protocol impossible;
* not using antihypertensive medication and using beta-blocker and/or alpha-blocker medication.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability. | 4 hours
  Analysis of heart rate variability with Wincardio Digital ECG.

CONTACTS AND LOCATIONS:
Locations (1):
- Diego Silveira da Silva, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No